CLINICAL TRIAL: NCT02843789
Title: Evolution of Adipokines and Body Composition in Rheumatoid Arthritis Patients Receiving Tocilizumab Therapy
Acronym: ADIPRAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2011/118
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: Adipokines; Tocilizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adiponectin evaluation (Experimental): Patients evaluated for serum adiponectin level and for body composition before each infusion of Tocilizumab
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab

SUMMARY:
The aim of this study is to analyze the variation of adiponectinemia and its molecular forms in RA patients receiving tocilizumab therapy.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease associated with cardiovascular morbidity. Tocilizumab (TCZ), a monoclonal antibody against the interleukin-6 receptor is an effective new biotherapy for the treatment of RA. This treatment is associated with increased LDL and HDL-cholesterol lipid parameters. Adipokines are adipose tissue-specific secreted molecules, which have many functions such as regulation of appetite, blood glucose or immune response. Among the adipokines, adiponectin exerts beneficial effects on the cardiovascular system. Patients with RA also exhibit body composition changes, including an increase in abdominal visceral fat. The impact of tocilizumab therapy in RA patients on adipokines and body composition is not known.

This project aims to explore the evolution of circulating adiponectin and other adipokines during tocilizumab therapy in RA. Body composition and its variations under tocilizumab therapy will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of RA and requiring Tocilizumab therapy
* Subject has provided written informed consent

Exclusion Criteria:

* Corticosteroid therapy (10 mg/day of prednisone or equivalent)
* Pregnant or lactating women
* Uncontrolled type 1 or type 2 diabetes
* Uncontrolled dyslipidemia
* Elevated transaminases (> three times higher than the normal range)
* History of diverticulitis or intestinal perforation
* Tocilizumab contraindications: Severe or active infections, Hypersensitivity to the active substance or to any of the excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Serum total adiponectin (ng/ml) | 12 months

SECONDARY OUTCOMES:
Serum high-molecular weight adiponectin (ng/ml) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Toussirot, Professor, Principal Investigator — University Hospital, Besançon, France
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toussirot E, Marotte H, Mulleman D, Cormier G, Coury F, Gaudin P, Dernis E, Bonnet C, Damade R, Grauer JL, Abdesselam TA, Guillibert-Karras C, Liote F, Hilliquin P, Sacchi A, Wendling D, Le Goff B, Puyraveau M, Dumoulin G. Increased high molecular weight adiponectin and lean mass during tocilizumab treatment in patients with rheumatoid arthritis: a 12-month multicentre study. Arthritis Res Ther. 2020 Sep 29;22(1):224. doi: 10.1186/s13075-020-02297-7. PMID 32993784